CLINICAL TRIAL: NCT04013282
Title: Adrenergic Cholinergic Enteric Measures/Mapping
Acronym: ACEM
Status: Recruiting | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Thomas Abell, Professor, University of Louisville
Other Study IDs: 13.0020.02
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients seen who had autonomic and enteric profiling (Adrenergic, Cholinergic, Enteric Measures/Mapping=ACEM_ from 2012-2019 at the University of Louisville.

DETAILED DESCRIPTION:
1. Patients seen who had autonomic and enteric profiling (Adrenergic Cholinergic Enteric Measures/Mapping=ACEM) from 2012-2019 at the U of Louisville.
2. Results of the physiologic measures of ACEM had the results recorded.
3. ACEM is compared to standardized gastric emptying values as the primary measure.
4. ACEM is also compared to metabolic measures of weight, height and thus BMI as a secondary measure.
5. ACEM is aloes compared with standardized gastrointestinal symptoms by a traditional patient recorded outcome as another secondary measure.

Other sites may be added if they have identical IRB and/or data sharing agreements with the University of Louisville.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the symptoms suggestive of autonomic and/or enteric disorders.

Exclusion Criteria:

* Anatomic obstruction of the GI tract
* Pregnancy
* Inability of patient or guardian to sign informed consent, if needed
* Psychiatric disorders precluding assessment and treatment of the patient's GI condition.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients seen
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-10-01; Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | 10 years
  We calculate Body Mass Index (BMI) using the following formula:
  weight (kg) / [height (m)] squared
  BMI is weight in kilograms divided by height in meters squared.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Abell, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States